CLINICAL TRIAL: NCT06908031
Title: Short-Course Radiotherapy Combined With mFOLFOX6, PD-1 Antibody and Cetuximab (for RAS/BRAF Wild-Type)/Bevacizumab (for RAS/BRAF Mutant) in High-Risk pMMR/MSS Rectal Adenocarcinoma: a Prospective, Multicenter Phase II Study
Brief Title: SCRT + mFOLFOX6 + PD-1 Antibody + Targeted Therapy for HIgh-Risk pMMR/MSS Rectal Cancer
Acronym: CRIT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jun Huang, Professor, Sixth Affiliated Hospital, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E2025076
Record Dates: First submitted 2025-04-01; First posted 2025-04-03 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-04

CONDITIONS: Rectal Adenocarcinoma; High-Risk Cancer; MSS
Keywords: Short-Course Radiotherapy; Targeting Therapy; Immunotherapy
MeSH Terms: conditions — Rectal Neoplasms | interventions — spartalizumab; Cetuximab; Bevacizumab; Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: The neoadjuvant treatment phase includes short-course radiotherapy (SCRT) combined with four cycles of the mFOLFOX6 regimen, PD-1 monoclonal antibody, and molecularly targeted drugs (selected based on RAS status; patients with RAS/BRAF wild-type receive cetuximab, while those with RAS/BRAF mutations receive bevacizumab). After completing the first cycle of mFOLFOX6 chemotherapy combined with targeted and immune therapy, patients undergo SCRT at a dose of 5Gy × 5 fractions. At least 7 days after the completion of radiotherapy, patients continue with three additional cycles of mFOLFOX6 chemotherapy combined with PD-1 monoclonal antibody and targeted drugs (bevacizumab is not used in the last cycle of the bevacizumab group). Surgery is performed 8-10 weeks after the completion of SCRT
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SCRT + mFOLFOX6 + PD-1 Antibody + Targeted Therapy (Experimental): The neoadjuvant treatment phase includes short-course radiotherapy (SCRT) combined with four cycles of the mFOLFOX6 regimen, PD-1 monoclonal antibody, and molecularly targeted drugs (selected based on RAS status; patients with RAS/BRAF wild-type receive cetuximab, while those with RAS/BRAF mutations receive bevacizumab). After completing the first cycle of mFOLFOX6 chemotherapy combined with targeted and immune therapy, patients undergo SCRT at a dose of 5Gy × 5 fractions. At least 7 days after the completion of radiotherapy, patients continue with three additional cycles of mFOLFOX6 chemotherapy combined with PD-1 monoclonal antibody and targeted drugs (bevacizumab is not used in the last cycle of the bevacizumab group). Surgery is performed 8-10 weeks after the completion of SCRT.
  Interventions: Radiation: Short-Course Radiotherapy; Drug: PD-1 monoclonal antibody; Drug: mFOLFOX6 regimen; Drug: Cetuximab; Drug: Bevacizumab; Procedure: Surgical resection

INTERVENTIONS:
Radiation: Short-Course Radiotherapy — Patients undergo SCRT at a dose of 5Gy × 5 fractions
  Other Names: SCRT
Drug: PD-1 monoclonal antibody — Patients complete immune therapy with PD-1 monoclonal antibody for 4 cycles.
  Other Names: PD-1
Drug: mFOLFOX6 regimen — Patients complete chemotherapy with mFOLFOX6 regimen for 4 cycles.
  Other Names: mFOLFOX6
Drug: Cetuximab — Patients with RAS/BRAF wild-type receive targeting therapy with Cetuximab for 4 cycles.
  Other Names: Cetuximab Antibody
Drug: Bevacizumab — Patients with RAS/BRAF mutations receive targeting therapy with Bevacizumab for 3 cycles. (Bevacizumab is not used in the last cycle of the bevacizumab group)
  Other Names: Bevacizumab Antibody
Procedure: Surgical resection — Surgery either local excition or total mesorectal excision is performed 8-10 weeks after the completion of short-course radiotherapy.
  Other Names: Surgery

SUMMARY:
To explore the efficacy and safety of short-course radiotherapy combined with mFOLFOX6, PD-1 monoclonal antibody and cetuximab (for RAS/BRAF Wild-Type)/bevacizumab (for RAS/BRAF Mutant) in High-Risk pMMR/MSS Rectal Adenocarcinoma through a prospective study, providing high-level evidence-based medical evidence for the use in the treatment of high-risk rectal cancer.

DETAILED DESCRIPTION:
Patients with locally advanced rectal cancer (LARC) who have high-risk factors, such as low rectal cancer, clinical stage T4b, positive mesorectal fascia (MRF), and positive extramural vascular invasion (EMVI), are at extremely high risk of distant metastasis. For these LARC patients with high-risk factors, the pathological complete response (PCR) rate with neoadjuvant chemotherapy alone is relatively low, ranging from 4.3% to 13.3%. Therefore, the use of a more potent comprehensive neoadjuvant treatment regimen, including concurrent chemoradiotherapy combined with targeted therapy and immunotherapy, may offer greater benefits to these patients. For patients with high-risk LARC, this study aims to explore whether the combination of short-course radiotherapy, mFOLFOX6, PD-1 monoclonal antibody and cetuximab (for RAS/BRAF Wild-Type)/bevacizumab (for RAS/BRAF Mutant) can improve the pathological responce rate, and achieve better long-term survival benefits. The study will investigate the efficacy and safety of short-course radiotherapy, mFOLFOX6, PD-1 monoclonal antibody and cetuximab (for RAS/BRAF Wild-Type)/bevacizumab (for RAS/BRAF Mutant) for high-risk LARC in treating liver metastases, with the goal of providing high-level evidence-based medical evidence for the use of local hypofractionated radiotherapy combined with PD-1 monoclonal antibody in the treatment of unresectable colorectal cancer liver metastasis.

This is a prospective, open-label, multicenter, single-arm, Phase II study. Patients with high-risk LARC will be eligible for enrollment.

Enrolled patients will receive neoadjuvant treatment phase includes short-course radiotherapy (SCRT) combined with four cycles of the mFOLFOX6 regimen, PD-1 monoclonal antibody, and molecularly targeted drugs (selected based on RAS status; patients with RAS/BRAF wild-type receive cetuximab, while those with RAS/BRAF mutations receive bevacizumab). After completing the first cycle of mFOLFOX6 chemotherapy combined with targeted and immune therapy, patients undergo SCRT at a dose of 5Gy × 5 fractions. At least 7 days after the completion of radiotherapy, patients continue with three additional cycles of mFOLFOX6 chemotherapy combined with PD-1 monoclonal antibody and targeted drugs (bevacizumab is not used in the last cycle of the bevacizumab group). Surgery is performed 8-10 weeks after the completion of SCRT. If pelvic MRI indicates clinical complete response (CCR) and N0, local excision (local excision, LE) will be performed. If pelvic MRI suggests clinical restaging as T1N0M0, LE surgery will be carried out. Otherwise, total mesorectal excision (TME) will be performed. The decision regarding adjuvant chemotherapy after surgery will be made by the attending physician.

ELIGIBILITY:
Inclusion Criteria:

1. Before conducting procedures related to the research protocol but not part of routine care, written informed consent, voluntarily signed and dated by the subject, must be obtained in accordance with regulations and institutional guidelines.
2. Age 18-75 years.
3. Histologically or cytologically confirmed pMMR/MSS rectal adenocarcinoma; all other histological types are excluded.
4. Distance from the lower margin of the rectal tumor to the anal verge ≤10 cm.
5. Clinical staging with high-risk factors, including cT3Nx, EMVI(+), or cT4, ±MRF(+), ±EMVI(+).
6. No evidence of distant metastasis before treatment.
7. No prior anti-cancer treatment (radiotherapy, chemotherapy, targeted therapy, or immunotherapy).
8. ECOG performance status of 0-1.
9. Peripheral blood counts and liver and kidney function within the following allowable ranges (tested within 15 days before the start of treatment):

   1. White blood cells (WBC) ≥3.0×10^9/L or absolute neutrophil count (ANC) ≥1.5×10^9/L;
   2. Hemoglobin (HGB) ≥80 g/L;
   3. Platelets (PLT) ≥100×10^9/L;
   4. Liver transaminases (AST/ALT) <3.0 times the upper limit of the normal range;
   5. Total bilirubin (TBIL) <1.5 times the upper limit of the normal range;
   6. Creatinine (CREAT) <1.5 times the upper limit of the normal range.
10. No history of other malignancies; not pregnant or breastfeeding, and effective contraception must be used during the study period and for 6 months after the last dose.

Exclusion Criteria:

1. Patients with a history of severe drug allergies (including allergies to platinum agents, 5-FU, LV, and 5-HT3 receptor antagonists);
2. Patients who have participated in or are currently participating in other clinical trials within 4 weeks prior to enrollment;
3. A history of having received anti-PD-1, PD-L1, PD-L2, CTLA-4, or any other specific T-cell costimulatory or checkpoint pathway-targeted therapy;
4. Severe electrolyte abnormalities;
5. Presence of gastrointestinal diseases, such as active ulcers in the stomach or duodenum, ulcerative colitis, or tumors with active bleeding that have not been resected; or other conditions that may lead to gastrointestinal bleeding or perforation; or gastrointestinal perforation that has not healed after surgical treatment;
6. History of arterial thrombosis or deep vein thrombosis within 6 months; history of bleeding or evidence of bleeding tendency within 2 months; or patients receiving high-dose anticoagulation therapy;
7. Pregnant or breastfeeding women, or women of childbearing potential with a positive pregnancy test before the first dose; or female participants and their partners who are unwilling to strictly practice contraception during the study period;
8. Presence of other active malignancies (except for malignancies that have been treated with curative intent and have been disease-free for more than 3 years, or in situ cancers that can be cured with adequate treatment);
9. Presence of severe ECG abnormalities or active coronary artery disease, severe/unstable angina, newly diagnosed angina or myocardial infarction within 12 months prior to study entry, or New York Heart Association (NYHA) Class II or higher congestive heart failure;
10. Patients with active infections (infections causing fever above 38°C);
11. Patients with uncontrolled hypercalcemia, hypertension, or diabetes;
12. Patients with severe pulmonary diseases (interstitial pneumonia, pulmonary fibrosis, severe emphysema, etc.);
13. Patients with psychiatric disorders that may affect clinical treatment or a history of central nervous system diseases;
14. Patients with severe complications (bowel obstruction, renal insufficiency, hepatic insufficiency, cerebrovascular disorders, etc.);
15. Presence of any CTCAE Grade 2 or higher toxicity caused by previous treatments that has not resolved (excluding anemia, alopecia, and skin pigmentation);
16. Any unstable medical condition that may affect patient safety and compliance with the study;
17. Patients deemed by the investigator as unsuitable for participation in this clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2025-04-02 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
pCR rate | 1 year
  pathological complete response rate

SECONDARY OUTCOMES:
3 years DFS Rate | 3 years
  3 years Disease Free Survival Rate
3 years OS rate | 3 years
  3 years Overall Survival Rate
3 years DMFS Rate | 3 years
  3 years Disease Metastasis Free Survival Rate
3 years RFS Rate | 3 years
  3 years Recurrence Free Survival Rate
R0 resection rate | 1 year
  R0 resection rate in participants
Toxicities Associated with Neoadjuvant Therapy | 1 year
  Incidence of adverse events related to neoadjuvant therapy as assessed by CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Juan Huang, PhD., Principal Investigator — Sun Yat-sen University
Locations (1):
- Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China